CLINICAL TRIAL: NCT03801460
Title: Physiological Reconditioning Program Administered Remotely in Patients Undergoing Transcatheter Aortic Valve Replacement Pilot Study
Brief Title: Physiological Reconditioning Program Administered Remotely in Patients Undergoing Transcatheter Aortic Valve Replacement: A Pilot Study
Acronym: PREPARE-TAVR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC201810
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Frailty; Transcatheter Aortic Valve Replacement; Rehabilitation
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized trial with objective end points assessment
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessed in a blinded manner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC (No Intervention): Standard of Care
- RAPR (Experimental): Remotely administered physiological reconditioning program
  Interventions: Other: Remotely administered physiological reconditioning program

INTERVENTIONS:
Other: Remotely administered physiological reconditioning program — Patients assigned to intervention arm will be provided a personalized, tailored and graduated exercise program to improve physical strength and conditioning.
  Arms: RAPR

SUMMARY:
The PREPARE TAVR pilot study will examine the effects of remotely administered physiological reconditioning program (RAPR) on quality of life (QOL) and clinical outcomes at one year post TAVR in frail older adults.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the effects of a home based exercise and dietary intervention program on the quality of life (QOL) and clinical outcomes in frail adults undergoing Transcatheter aortic valve replacement (TAVR) procedures. Patients will be randomly (1:1) assigned to the standard of care (SOC group) where patients will receive all medical care as decided by their treating physicians or assigned to a home based program known as remotely administered physiological reconditioning (RPR) program which will include receiving personalized instructions for a progressive exercise program and dietary changes. Patients will be contacted for regular phone and in-person follow up for monitoring their progress. The primary endpoint will be quality of life as assessed by KCCQE questionnaires at one-year post TAVR. The secondary endpoints include length of stay post TAVR, all-cause mortality, repeat hospitalization and a composite of all-cause mortality and repeat hospitalization at one year.

ELIGIBILITY:
Inclusion Criteria:

- Short Physical Performance Battery Protocol (SPPB) score < 9

Exclusion Criteria:

* Severe liver disease defined by Childs Pugh class >B or MELD score >15.
* Severe kidney disease defined by eGFR <30 mL/min.
* Hospital admission during the 4 weeks prior to randomization.
* Montreal objective cognitive assessment (MOCA) score <18.
* Mechanical fall in the past month.
* Unstable angina during the previous month.
* Myocardial infarction during the previous month.
* Unsuccessful completion of the one-week run-in phase.
* Syncopal episode during exercise during run-in phase

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QOL) | One year
  Quality of life as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ). KCCQE is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life (QOL) within a 2-week recall period. KCCQ responses are provided along a rating scale continuum with equal spacing from worst to best.

SECONDARY OUTCOMES:
LOS | Index hospitalization
  Length of stay post TAVR
MACE | one year
  Composite of mortality and repeat hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Asim Cheema, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- Southlake Hospital, Newmarket, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abraham LN, Sibilitz KL, Berg SK, Tang LH, Risom SS, Lindschou J, Taylor RS, Borregaard B, Zwisler AD. Exercise-based cardiac rehabilitation for adults after heart valve surgery. Cochrane Database Syst Rev. 2021 May 7;5(5):CD010876. doi: 10.1002/14651858.CD010876.pub3. PMID 33962483